CLINICAL TRIAL: NCT03903887
Title: A Phase I/II Study of Combination of Anti-Programmed Cell Death Protein1 (Anti-PD1) Antibody-activated Autologous Tumor Infiltrating Lymphocytes (TILs) and Chemotherapy in the Treatment of Stage II-IIIA Non-small Cell Lung Cancer
Brief Title: A Study of Anti-PD1 Antibody-activated TILs in Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jianchuan Xia, Director of Biotherapy, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2018-149-02
Record Dates: First submitted 2019-03-31; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung Cancer; TIL; immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD1-TIL combined with chemotherapy (Experimental): Participants would receive anti-PD1 antibody-activated TILs after the final cycle of adjuvant chemotherapy.
  Interventions: Biological: anti-PD1 antibody-activated TILs

INTERVENTIONS:
Biological: anti-PD1 antibody-activated TILs — Participants would receive one dose of anti-PD1 antibody-activated TILs at the final cycle of docetaxel and cisplatin (DP) regimen chemotherapy.

SUMMARY:
This study was a phase I/II trial initiated by the investigator to evaluate the safety and tolerability of anti-PD-1 antibody-activated TILs combined with adjuvant chemotherapy in participants with stage II-IIIA non-small cell lung cancer. 20 participants were enrolled and anti-PD-1 antibody-activated TILs was infused into participants after the final cycle chemotherapy to assess the safety and disease-free survival.

DETAILED DESCRIPTION:
Postoperative non-small cell lung cancer received 4 cycles of docetaxel and cisplatin regimen adjuvant chemotherapy and received anti-PD1 antibody-activated TILs on the day 15 of the final cycle of chemotherapy.

Fresh tumor tissues or sentinel lymph nodes were collected from participants with postoperative non-small cell lung cancer, and the tumor tissues were digested with type IV collagenase at 37 °C for 2 to 4 hours. The cell pellet was washed, suspended in medium containing 10% AB serum, planted in a 24-well cell culture plate, and periodically changed according to the growth of the cells. After culturing for 2 to 3 weeks, TILs were co-stimulated with radioactively irradiated allogeneic peripheral blood mononuclear cells （PBMCs）and were expanded in 100 ml of Interleukin-2 (IL-2) medium in a cell culture flask. After rapid expansion for 15 days, the number of cells reached 0.1-1*10^10 cells. Before cell transfer, TILs were incubated with anti-PD-1 antibody, and a fraction of the TILs were collected to assess their number, phenotype, and viability of cells, and to test for possible contamination by bacteria, fungi, or endotoxins. Then, autologous TILs (0.1-1*10^10 cells) were transferred to participants via intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

* Participants with stage II-IIIA non-small cell lung cancer and scheduled to receive adjuvant chemotherapy postoperation.
* Age 18 to 75 years.
* Willing to sign a durable power of attorney.
* Able to understand and sign the Informed Consent Document.
* Life expectancy of greater than six months.
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after receiving the preparative regimen.
* Adequate organ function.
* Serology:

Seronegative for HIV antibody. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.

* Hematology:

white blood cell count (> 3500/mm(3)). Platelet count greater than 100,000/mm(3). Hemoglobin greater than 9.0 g/dl.

* Chemistry:

Serum Alanine aminotransferase/Aspartate aminotransferase less or equal to 2.5 times the upper limit of normal.

Serum creatinine less than or equal to 1.6 mg/dl. Total bilirubin less than or equal to 1.5 mg/dl.

Exclusion Criteria:

* Previous treatment with anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) , anti-PD-1, and anti-Programmed death-ligand 1(PD-L1).
* Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
* Allogeneic tissue/organ transplantation.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* History of autoimmune disease
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* Concurrent antineoplastic therapies and systemic steroid therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Severity of adverse events | 3 weeks
  According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE)

SECONDARY OUTCOMES:
Disease-free survival (DFS) | 6 months
  DFS is defined as the time from surgery until tumor recurrence or death.
Overall survival (OS) | 12 months
  OS is defined as the time from surgery until death from any cause
The quality of life by EQ-5D-5L (EuroQol Group, Chinese versions ) | 3 weeks
  Participants were interviewed with the EQ-5D-5L (EuroQol Group, Chinese versions). There are numbers from 0 to 100 on this scale of the EQ-5D-5L. 100 represents the best health condition you can imagine, and 0 represents the worst health condition in your imagination. Please put an X on the scale to indicate how healthy you are today. And the number you marked on the scale represents your health condition today.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen University, Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
We did not decide whether to share the subject's personal information.